CLINICAL TRIAL: NCT00002113
Title: A Pilot Study of Fluconazole Plus Flucytosine for the Treatment of AIDS Patients With Acute Cryptococcal Meningitis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pfizer (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 213A; R-0202
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1996-04

CONDITIONS: Meningitis, Cryptococcal; HIV Infections
Keywords: Meningitis; Cryptococcosis; Drug Therapy, Combination; Fluconazole; Flucytosine; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — Meningitis, Cryptococcal; HIV Infections; Meningitis; Cryptococcosis; Acquired Immunodeficiency Syndrome | interventions — Flucytosine; Fluconazole

INTERVENTIONS:
Drug: Flucytosine
Drug: Fluconazole

SUMMARY:
To evaluate and estimate the safety and efficacy of the combination of fluconazole and flucytosine as treatment for acute cryptococcal meningitis in patients with AIDS.

Fluconazole and flucytosine have different mechanisms of action. Since fluconazole has not been associated with hematologic suppression and does not produce renal impairment that can result in higher serum flucytosine levels, this combination may be better tolerated than is amphotericin B plus flucytosine.

DETAILED DESCRIPTION:
Fluconazole and flucytosine have different mechanisms of action. Since fluconazole has not been associated with hematologic suppression and does not produce renal impairment that can result in higher serum flucytosine levels, this combination may be better tolerated than is amphotericin B plus flucytosine.

Patients in each cohort receive a lower dose of fluconazole alone or in combination with flucytosine, or a higher dose of fluconazole alone. Doses in subsequent cohorts are escalated if safety data in the previous cohort is satisfactory. Patients are evaluated weekly for the first 4 weeks and every 2 weeks thereafter. Therapy continues until 8 weeks after the CSF becomes culture negative, up to a maximum of 26 weeks.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Antiviral therapy (AZT, DHPG).
* Prophylaxis for Pneumocystis carinii pneumonia.
* Treatment for intercurrent opportunistic infection.

Concurrent Treatment:

Allowed:

* Radiation therapy for mucocutaneous Kaposi's sarcoma.

Patients must have:

* AIDS.
* Evidence of Cryptococcal neoformans in culture or lumbar CSF OR clinical and CSF findings compatible with cryptococcal meningitis.
* No evidence of acute or chronic meningitis of any etiology other than cryptococcosis.
* Life expectancy of at least 2 weeks.

Prior Medication:

Allowed:

* Prior antiviral therapy (AZT, DHPG).
* Prophylaxis for Pneumocystis carinii pneumonia.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Relapsing on maintenance triazole therapy for cryptococcal meningitis.
* Unable to take oral medication.

Concurrent Medication:

Excluded:

* Concomitant use of any antifungal agent other than study drug.

Patients with the following prior conditions are excluded:

History of allergy to or intolerance of imidazoles, azoles, or flucytosine.

Prior Medication:

Excluded:

* More than 1 mg/kg amphotericin B.
* Systemic antifungal agents within 7 days prior to study entry.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Los Angeles County - USC Med Ctr, Los Angeles, California
  - UCI Med Ctr, Orange, California
  - UCSD Med Ctr - Owen Clinic, San Diego, California

REFERENCES:
- [Background] Larsen RA, Bozzette SA, Jones BE, Haghighat D, Leal MA, Forthal D, Bauer M, Tilles JG, McCutchan JA, Leedom JM. Fluconazole combined with flucytosine for treatment of cryptococcal meningitis in patients with AIDS. Clin Infect Dis. 1994 Oct;19(4):741-5. doi: 10.1093/clinids/19.4.741. PMID 7803641